CLINICAL TRIAL: NCT02748668
Title: Extracorporeal Membrane Oxygenation: Blood Cells
Brief Title: Extracorporeal Membrane Oxygenation (ECMO): Blood Cells
Status: Terminated | Type: Observational
Why Stopped: Study was not able to achieve primary objective and there is no intention to work towards its achievement
Sponsor: Corewell Health West (Other)
Collaborators: Van Andel Research Institute (Other)
Responsible Party: Principal Investigator, Renzo Loyaga Rendon, Medical Director of Cardiovascular Research, Corewell Health West
Other Study IDs: 2014-255
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Extracorporeal Membrane Oxygenation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Days
Biospecimen Retention: Samples Without DNA — Blood is collected for analysis of cytokines and inflammatory cell patterns, and will be stored for future research.

GROUPS / COHORTS (2):
- ECMO: No intervention. Blood specimen collection.
  Interventions: Other: Blood specimen collection
- Control: No intervention. Blood specimen collection.
  Interventions: Other: Blood specimen collection

INTERVENTIONS:
Other: Blood specimen collection

SUMMARY:
The objective of the study is to predict outcomes of patients on extracorporeal membrane oxygenation (ECMO) therapy by correlating cytokines and inflammatory cell patterns to clinical outcomes using data collected in the ECMO Registry at Spectrum Health.

ELIGIBILITY:
ECMO group:

Inclusion Criteria:

* Greater than or equal to 18 years of age
* Subject presents to the CTICU at Butterworth Campus, Spectrum Health and is critically ill in the ICU needing ECMO therapy.

Exclusion Criteria:

* Subject is less than 18 years of age
* Known prisoner

Control Subjects:

Inclusion Criteria

* Greater than 18 years of age
* Without any known cardiovascular, lung, or autoimmune disease.

Exclusion Criteria:

* Less than or equal to 18 years of age
* Known cardiovascular, lung, or autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients on ECMO and 100 control patients will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Renzo Loyaga-Rendon, MD,PhD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States